CLINICAL TRIAL: NCT02014987
Title: The Initial Running Volume and Running Related Injury Among Novice Runners
Brief Title: Running Related Injury Among Novice Runners
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: N-20130035
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Treatment Error; Overuse Injury
Keywords: Running related injury; Overuse injury; Running pattern
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Running training programmes (Experimental): Runners with a high body mass index are going to follow a training programme of 3 kilometres per week compared to a training programme of 6 kilometres per week.
  The amount of running will be increased with 10 % per week.
  Interventions: Behavioral: Training programmes

INTERVENTIONS:
Behavioral: Training programmes — Runners with a high body mass index follow two types of training programmes:
  1. a running programme of 3 kilometres per week
  2. a running programme 6 kilometres per week
  The amount of running will be increased with 10 % per week.

SUMMARY:
About 31% of the Danish population participates regularly in running. The positive health benefits of running have been well documented in the literature. Unfortunately, running has been connected with a high risk of injuries.

Running related injuries can cause a long rehabilitation and may even force the runner to quit running permanently. To ensure that running can be practiced as a safe exercise activity prevention must be considered.

DETAILED DESCRIPTION:
Training errors (i.e. excessive volume, sudden change of training routines etc.) are held to be the main reasons to running related injuries. Fortunately, training errors can be avoided as training characteristics (distance, duration, pace) can be controlled by the runner.

In order to avoiding training errors, especially excessive volume many novice runners follow 0-5 kilometres type training programmes. However, limited research has been conducted on the training volume of beginner programs and the risk of running related injuries.

The purpose of this study is to investigate the relationship between the running volume the first 4 weeks of a running regime and the risk of running related injuries among novice runners. The relationship between running volume and running related injuries will be investigated in proportion to their body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* both gender between 16-65 years
* no running-training within the last year
* less than 20 hours of sports activity within the last year (in total)
* internet access and mail address
* body mass index between 18.5 - 25 or 30-35
* owns a pair of running shoes

Exclusion Criteria:

* do not want to use a GPS watch
* unable or unwilling to follow the running regime in 4 consecutive weeks
* previous injury in lower extremity within the last 2 years
* unable to read or understand Danish
* former heart surgery
* known heart surgery
* known lung disease
* diabetes
* current pregnancy
* known tendency to shortness of breath or chest pain with activity
* known tendency to leg pain when walking long distances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Running related injury | 7 days
  An injury sustained on muscles, joints, tendons and/or bones during or after running. The injury must have caused a workout reduction (reduced distance, intensity, frequency etc.) for at least 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Bertelsen, PT, Study Chair — Department of Publich Health, Aarhus University; Sten Rasmussen, MD, Principal Investigator — Northern Orthopaedic Division, Aalborg University Hospital
Locations (1):
- Sten Rasmussen, Aalborg, Northern Jutland, Denmark